CLINICAL TRIAL: NCT04828707
Title: A Prospective, Randomized, Double-blind, Sham-controlled Multi-center Clinical Study Assessing the Safety and Efficacy of Nerivio for the Preventive Treatment of Migraine
Brief Title: Assessment of Safety and Efficacy of Nerivio for the Migraine Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theranica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TCH008
Record Dates: First submitted 2021-03-30; First posted 2021-04-02 (Actual); Results first posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2022-03

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, sham-controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Migraine prevention treatment with active Nerivio (Active Comparator): Participants will treat with an active Nerivio device every other day for migraine prevention.
  Interventions: Device: Nerivio active device
- Migraine prevention treatment with sham Nerivio (Sham Comparator): Participants will treat with a sham (placebo) Nerivio device every other day for migraine prevention.
  Interventions: Device: Nerivio sham device

INTERVENTIONS:
Device: Nerivio active device — Nerivio neurostimulator of conditional pain modulation (CPM)
  Arms: Migraine prevention treatment with active Nerivio
Device: Nerivio sham device — Nerivio neurostimulator with an electrical output not intended for neurostimulation
  Arms: Migraine prevention treatment with sham Nerivio

SUMMARY:
Migraine is a common neurologic with attacks of headache and associated symptoms such as nausea, vomiting, phono and photophobia. Migraine can lead to substantial functional impairment. This study intends to demonstrate the safety and efficacy of the Nerivio for migraine prevention.

The study is a prospective, randomized, double-blind, sham-controlled, multicenter study, conducted in three phases.

The study will consist of a screening/enrollment visit, followed by a 4-week (28 days) baseline phase, an 8-week double-blind preventive treatment phase, and a 4-week open-label phase.

Patients will complete an electronic diary throughout the study; this includes a daily evening report (completed regardless of whether the patient had a headache) and treatment feedback during the follow-up pre-emptive phase.

The primary endpoint is the mean change in the average of migraine headache days per month comparing the 4-week baseline phase (weeks 1 through 4) with the last 28 days of the treatment phase (weeks 9 through 12).

DETAILED DESCRIPTION:
Nerivio is a neuromodulation device approved for the acute treatment of migraine with or without aura in patients 12 years of age or older. The device utilizes electro stimulation to achieve conditioned pain modulation (CPM). CPM stimulate endogenous analgesic mechanism. Treatments are self-administered by the user at the onset of a migraine attack. this study intends to demonstrate the safety and efficacy of the Nwrivio for migraine prevention.

The study is a prospective, randomized, double-blind, sham-controlled, multicenter trial, conducted in three phases. The ratio between treatment and control groups will be 1:1, stratified by center and patient type (chronic/non-chronic). The study will consist of a screening/enrollment visit, followed by a 4-week (28 days) baseline phase. Eligible participants will enter an 8-week double-blind preventive treatment phase. Following the preventive treatment phase, patients will be offered to participate in a 4-week open-label pre-emptive treatment phase or continue their prevention treatment with an active device, according to their eligibility.

Patients will complete an electronic diary throughout the study; this includes a daily evening report (completed regardless of whether the patient had a headache) and treatment feedback during the follow up pre-emptive phase

Phase I - Baseline - 4 weeks (weeks 1 through 4):

Eligible participants will install the Nerivio app on their smartphones and will be instructed to record daily their migraine/headaches symptoms and medication use on the Nerivio app.

Transition to the treatment phase: Participants who meet the following criteria in the baseline phase will be eligible to continue to the treatment phase:

* Complete the diary in at least 22 out of the 28 days during the baseline phase (80%)
* Have between 6 to 24 headache days during the 28-day baseline period
* At least 4 of their headache days during the baseline phase fulfill the International Classification of Headache Disorders 3rd edition (ICHD-3) criteria for migraine (migraine without aura [code 1.1; C and D] or with aura [code 1.2; B and C], or probable migraine, or headaches requiring the use of migraine-specific medications including triptans, gepants or ergot derivatives).

Phase II - treatment phase (prevention) - 8 weeks (weeks 5 through 12):

Participants who meet the baseline phase requirements will be randomized in a 1:1 ratio to active and sham groups. Participants will be instructed to complete a daily diary (in the Nerivio app) about their headaches, associated symptoms, and medication use. They will also be instructed to conduct a 45-minute treatment with Nerivio every other day.

Transition to the follow-up phase (open label):

At the end of the treatment phase, participants from both arms (active and sham) may continue to a follow-up phase in which they will receive an active device that can be used during this phase. The data of all participants will be used for safety analyses.

The data of participants from the baseline and treatment phases will be used to assess their eligibility to participate in the pre-emptive follow-up phase. Participants eligible for the follow-up phase meet the following conditions:

* Between 6-16 headache days during the baseline phase.
* Participants experience prodrome symptoms within 24 hours prior to the onset of their migraine headache in at least half of their migraine attacks during the baseline phase.
* Participants completed the daily questionnaires in at least 70% of the days during the treatment phase.
* Treated every other day in at least 24 and less than 33 days during the 56 days of the treatment phase.

All adverse events will be reported.

Phase III - Follow-up phase (open label) - 4 weeks (weeks 13 through 16):

All participants will receive an active Nerivio device to use during the follow-up phase. Participants who do not meet the above requirements will be able to enter into the safety follow-up and continue to use Nerivio every other day for the preventive treatment of migraine. They will be instructed to compete a daily diary as was done in the treatment phase.

Participants who meet the above requirements will enter the pre-emptive follow-up phase and be instructed to conduct a 45-minute device treatment within 60 minutes of prodrome symptom onset. Participants will be instructed to complete questionnaires regarding their headache, prodrome symptoms, and medication use at baseline (start of treatment), 2 hours post-treatment, and 24 hours post-treatment. In addition, participants will be instructed to continue to report the daily diary, as performed in the other phases of the study.

All adverse events will be reported.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old.
2. Must have at least a 6-month history of headaches that meet the ICHD-3 diagnostic criteria for migraine with or without aura, either chronic (at least 15 days of Headache Days(HD)/ month with migraine days (migraine with or without aura) at least 8 days/ month for > 3 months) or non-chronic migraine.
3. History of 6 to 24 headache days per 28-day period for each of the 3 months preceding study enrolment (based on participant report).
4. Subject on prophylactic migraine treatment are permitted to remain on 1 medication with possible migraine-prophylactic effects if the dose has been stable for at least 2 months prior to the screening visit, and the dose is not expected to change during the course of the study.
5. Have personal access to a smartphone (24/7).
6. Must be able and willing to comply with the protocol.
7. Must be able and willing to provide informed consent..

Exclusion Criteria:

1. An active implanted electrical and/or neurostimulator device (e.g. cardiac pacemaker, cochlear implant).
2. Uncontrolled epilepsy.
3. History of use of opioids or barbiturates on more than 4 days a month in the last 6 months.
4. Current participation in any other interventional clinical study
5. Subject without basic cognitive and motor skills required for operating a smartphone.
6. Pregnant or breastfeeding.
7. Other significant pain, medical or psychological problems that in the opinion of the investigator may confound the study assessments.
8. Prior experience with the Nerivio device.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cowan, MD, Study Chair — Stanford Health Care
Locations (16):
- United States (16):
  - Evolve Clinical Research, Phoenix, Arizona
  - The Neurology Center of Southern California, Carlsbad, California
  - Newport Beach Clinical Research Associates, Newport Beach, California
  - Hartford Headache Center, Hartford, Connecticut
  - RecioMed Clinical Research, Boynton Beach, Florida
  - Beautiful Minds Clinical Research Center, Cutler Bay, Florida
  - Chicago Headache Center and Research Institute, Chicago, Illinois
  - Deaconess Clinic, Evansville, Indiana
  - Four Rivers Clinical Research, Paducah, Kentucky
  - Headache Neurology Research Institute, Ridgeland, Mississippi
  - StudyMetrix Research, City of Saint Peters, Missouri
  - ClinVest Research, Springfield, Missouri
  - Ocean medical research, Toms River, New Jersey
  - DENT Neurosciences Research Center, Amherst, New York
  - Prevention & Strengthening Solutions, Inc., Columbia, South Carolina
  - West Virginia University Medicine, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Monteith TS, Stark-Inbar A, Shmuely S, Harris D, Garas S, Ironi A, Kalika P, Irwin SL. Remote electrical neuromodulation (REN) wearable device for adolescents with migraine: a real-world study of high-frequency abortive treatment suggests preventive effects. Front Pain Res (Lausanne). 2023 Nov 6;4:1247313. doi: 10.3389/fpain.2023.1247313. eCollection 2023. PMID 38028429

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study contained a 4-week baseline phase, an 8-week treatment phase, and 4-week follow-up phase.
  Participants who had 6-24 headache days and completed at least 22 daily diaries at baseline were eligible to enter the treatment phase. out of the 335 recruited participants, 18 participants did not complete the baseline phase and 69 participants completed the baseline but were non-eligible to continue to the treatment phase. Thus, 248 participants were randomized into the treatment phase.
Groups:
- Migraine Prevention Treatment With Active Nerivio: Participants were treated with an active Nerivio device every other day for migraine prevention.
  Nerivio active device: Nerivio neurostimulator of conditional pain modulation (CPM)
- Migraine Prevention Treatment With Sham Nerivio: Participants were treated with a sham (placebo) Nerivio device every other day for migraine prevention.
  Nerivio sham device: Nerivio neurostimulator with an electrical output not intended for neurostimulation
Period: Overall Study
Arm/Group | Migraine Prevention Treatment With Active Nerivio | Migraine Prevention Treatment With Sham Nerivio
Started | 128 (248 out of the 335 enrolled participants were eligible for randomization following the baseline phase. out of these 248 participants, 128 were randomized into the Nerivio Active group) | 120 (248 out of the 335 enrolled participants were eligible for randomization following the baseline phase. out of these 248 participants, 120 were randomized into the Nerivio Sham group)
Completed | 123 | 117
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Migraine Prevention Treatment With Active Nerivio | Migraine Prevention Treatment With Sham Nerivio | Total
Number analyzed (Participants) | 128 | 120 | 248
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The analysis was performed on participants who completed the baseline phase and were randomized into the treatment groups
  years | 41.0 (12.0) | 42.6 (13.6) | 41.7 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 103 | 213
  Male | 18 | 17 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 9 | 15
  White | 116 | 106 | 222
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 128 | 120 | 248
Height [Mean (Standard Deviation); unit: cm] | 166 (8.4) | 165 (8.2) | 166 (8.3)
Weight [Mean (Standard Deviation); unit: Kg] | 84.0 (25.6) | 85.0 (25.2) | 84.5 (25.0)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.6 (8.3) | 31.2 (8.4) | 30.8 (7.7)

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Migraine Days
Description: The mean reduction in the number of migraine days per month during the last 28 days (4 weeks) of the treatment phase (weeks 9 through 12) compare to the 4-week baseline phase (weeks 1 through 4)
  A migraine day is defined as a calendar day with a headache that is accompanied by at least one of the following symptoms: aura, photophobia, phonophobia, nausea and/or vomiting; or a calendar day with a headache that is treated with a migraine-specific acute medication.
Time Frame: 3 months
Population: Participants who treated at least once with Nerivio device (either Active or Sham)
Measure: Mean (Standard Error); unit: Migraine days per month
Arm/Group | Migraine Prevention Treatment With Active Nerivio | Migraine Prevention Treatment With Sham Nerivio
Number analyzed (Participants) | 128 | 120
Migraine days per month | -3.8 (0.4) | -1.1 (0.4)
Statistical Analysis 1: Comparison: Migraine Prevention Treatment With Active Nerivio vs Migraine Prevention Treatment With Sham Nerivio; The Intent-To-Treat (ITT) dataset was used for primary outcome. To overcome impact of missing data, statistical analysis was conducted using the Last Observation Carried Forward (LOCF) as an imputation method. The data of each variable collected from the daily diary was normalized to 28 days for every period (weeks 1-4, weeks 5-8, and weeks 9-12). Participants' data who entered the treatment phase but dropped out during weeks 5-8 were carried forward and analyzed as their data at weeks 9-12; Test type: Superiority; p < 0.05, t-test, 2 sided

2. Primary Outcome: Rate of Adverse Events (Safety and Tolerability)
Description: Number of participants with Adverse Events (AE), Serious Adverse Events (SAE) and Device-related Adverse Events
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Migraine Prevention Treatment With Active Nerivio | Migraine Prevention Treatment With Sham Nerivio
Number analyzed (Participants) | 128 | 120
participants
  Adverse Events | 20 | 21
  Serious Adverse Events | 2 | 0
  Device related Adverse Events | 0 | 1
  Device related Serious Adverse Events | 0 | 0

3. Secondary Outcome: Reduction in Moderate/Severe Headache Days
Description: The mean reduction in the number of moderate/severe headache days per month during the last 28 days (4 weeks) of the treatment phase (weeks 9 through 12) compare to the 4-week baseline phase (weeks 1 through 4)
  A moderate/severe headache day is defined as a calendar day with a moderate or severe headache.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: Moderate/Severe headache days per month
Arm/Group | Migraine Prevention Treatment With Active Nerivio | Migraine Prevention Treatment With Sham Nerivio
Number analyzed (Participants) | 128 | 120
Moderate/Severe headache days per month | -3.5 (0.3) | -2.1 (0.4)

4. Secondary Outcome: Reduction Headache Days
Description: The mean reduction in the number of headache days per month during the last 28 days (4 weeks) of the treatment phase (weeks 9 through 12) compare to the 4-week baseline phase (weeks 1 through 4)
  A headache day is defined as a calendar day with headache (at any severity).
Time Frame: 3 months
Measure: Mean (Standard Error); unit: Headache days per month
Arm/Group | Migraine Prevention Treatment With Active Nerivio | Migraine Prevention Treatment With Sham Nerivio
Number analyzed (Participants) | 128 | 120
Headache days per month | -4.2 (0.4) | -2.0 (0.4)

5. Secondary Outcome: Reduction of 50% in Headache Days
Description: Percentage of patients achieving at least 50% reduction from baseline in the mean number of headache days (all severities) per month in the last 4 weeks of the treatment phase (weeks 9 through 12).
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Migraine Prevention Treatment With Active Nerivio | Migraine Prevention Treatment With Sham Nerivio
Number analyzed (Participants) | 128 | 120
Participants | 40 | 22

6. Secondary Outcome: Increase in Headache Impact Test-6 (HIT-6) Score at the End of the Last 28 Days (4 Weeks) of the Treatment Phase (Weeks 9 Through 12) Compare to the HIT-6 Score at the End of the 4-week Baseline Phase (Weeks 1 Through 4)
Description: Headache Impact Test-6 (HIT-6) questionnaire is a tool used to measure the impact headaches have on your ability to function on the job, at school, at home, and in social situations. the questionnaire contains 6 questions with a total score between 36 to 78. Higher score interpret as better patient outcome.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Migraine Prevention Treatment With Active Nerivio | Migraine Prevention Treatment With Sham Nerivio
Number analyzed (Participants) | 128 | 120
score on a scale | 4.7 (0.6) | 3.9 (0.6)

7. Secondary Outcome: Reduction in Migraine-Specific Quality-of-Life (MSQ) Questionnaire Score at the End of the Last 28 Days (4 Weeks) of the Treatment Phase (Weeks 9 Through 12) Compare to the MSQ Score at the End of the 4-week Baseline Phase (Weeks 1 Through 4)
Description: The migraine Specific Quality-of-Life questionnaire (MSQ) is a tool to measure the impact of migraine on your ability to function on the job, at school, at home, and in social situations. The questionnaire contains 14 questions with a total score between 0 to 84. Lower score interprets as better patient outcome.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Migraine Prevention Treatment With Active Nerivio | Migraine Prevention Treatment With Sham Nerivio
Number analyzed (Participants) | 128 | 120
score on a scale | -11.5 (1.1) | -9.8 (1.2)

8. Other Pre Specified Outcome: Reduction in Migraine Medication Intake
Description: Reduction in the mean number of acute headache/migraine medication days per month in the last 4 weeks of the treatment phase (weeks 9 through 12) compared to baseline (weeks 1 through 4).
Time Frame: 3 months
Measure: Mean (Standard Error); unit: Medication intake day per month
Arm/Group | Migraine Prevention Treatment With Active Nerivio | Migraine Prevention Treatment With Sham Nerivio
Number analyzed (Participants) | 128 | 120
Medication intake day per month | -3.9 (0.4) | -2.2 (0.4)

9. Other Pre Specified Outcome: Percentage of Freedom From Headache Post 2 Hours Following Prodrome Treatment
Description: Percentage of participants who treat for the first treatment in the pre-emptive phase, during the prodrome, when they are pain-free, and remain pain-free during the following 2 hours after the treatment, without use of acute medication.
Time Frame: 2 hours post treatment at follow up phase
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Percentage of Freedom From Headache Post 24 Hours Following Prodrome Treatment
Description: Percentage of participants who treat for the first treatment in the pre-emptive phase, during the prodrome, when they are pain-free, and remain pain-free during the following 24 hours after the treatment, without use of acute medication.
Time Frame: 24 hours post treatment at follow up phase
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Percentage of Reduction of Headache Post 24 Hours From Prodrome Treatment
Description: Percentage of patients who treat during the prodrome, when they are pain free, and remain either pain free or with mild pain during the following 24 hours after the treatment without use of acute medication.
Time Frame: 24 hours post treatment at follow up phase
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Feasibility of Migraine Prediction Algorithm
Description: Analysis of the daily information provided by the participants for the purpose of predicting their migraine days
Time Frame: 3 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Health Economic Analysis
Description: Health economics analysis of the difference between subjects using Nerivio as a therapy and those who do not with respect to:
  1. Absenteeism - number of missed work/school days
  2. Presenteeism - number of work/school days with moderate/severe functional disability
  3. Healthcare provider appointments
  4. ED visits
  5. Brain MRI/CT scans
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Migraine Prevention Treatment With Active Nerivio | Migraine Prevention Treatment With Sham Nerivio
All-Cause Mortality (participants affected / at risk) | 0/128 | 0/120
Serious Adverse Events (participants affected / at risk) | 2/128 | 0/120
Other Adverse Events (participants affected / at risk) | 20/128 | 21/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Migraine Prevention Treatment With Active Nerivio (N=128) | Migraine Prevention Treatment With Sham Nerivio (N=120)
SAE - suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) — Participant with stress/anxiety disorder tried to commit suicide during the treatment phase. The participant was hospitalized following the event and discontinued the study
SAE - falling in bathroom (Surgical and medical procedures) | 1 (1) | 0 (0) — The participant falls in the bathroom and hit his head on the sink. participant required medical treatment and decide to discontinue the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Migraine Prevention Treatment With Active Nerivio (N=128) | Migraine Prevention Treatment With Sham Nerivio (N=120)
COVID 19 (Infections and infestations) | 3 | 3
Sinusitis/common cold (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Bruises from falling (Musculoskeletal and connective tissue disorders) | 2 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Ear infection (Ear and labyrinth disorders) | 2 | 1
Migraine/headache worsening (Nervous system disorders) | 1 | 2
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 | 1
nfluenza (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dental Infection (Infections and infestations) | 1 | 0
Worsening of fibromyalgia pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Lipoma (Skin and subcutaneous tissue disorders) | 1 | 0
worsening of chronic rhinitis (Immune system disorders) | 0 | 1
cervical precancerous cells diagnosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Ankle fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Hornet Stings (Immune system disorders) | 1 | 0
Yeast infection (Infections and infestations) | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Worsening of Depression (Psychiatric disorders) | 0 | 1
Hyperlipidemia (Metabolism and nutrition disorders) | 1 | 0
Vaginal Itching (Reproductive system and breast disorders) | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 1
Overweight (Metabolism and nutrition disorders) | 0 | 1
Viral Infection (Infections and infestations) | 0 | 1

LIMITATIONS AND CAVEATS:
No limitations or caveats to report

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT04828707/Prot_SAP_001.pdf